CLINICAL TRIAL: NCT06157567
Title: Clinical Feasibility Study to Evaluate the Safety and Performance of the Profound Matrix System
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Candela Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PFX22003
Record Dates: First submitted 2023-11-16; First posted 2023-12-06 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Skin Laxity; Wrinkle; Skin Condition
MeSH Terms: conditions — Cutis Laxa; Skin Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Treatment Group (Experimental): Study subjects may be treated with any of the Profound Matrix applicators: Sublime, Sublative RF and/or Matrix Pro. Treatments may include combination of applicators or additional commercial devices per PI discretion.
  Interventions: Device: Profound Matrix

INTERVENTIONS:
Device: Profound Matrix — Treatment visits are limited to up to three (3) study treatments (with treatment intervals 6 weeks ± 2 weeks).

SUMMARY:
This is a non-randomized, multi-center, open-label clinical trial evaluating clinical feasibility treatments with the Profound Matrix system.

DETAILED DESCRIPTION:
The Profound Matrix system is a multipurpose (3-in-1) radiofrequency (RF) platform. The clinical study is to evaluate the safety and performance of the Profound Matrix system with Sublime applicator, RF applicator and Matrix Pro applicator for aesthetic treatments including its cleared indications of wrinkles, acne scars, striae, and electrocoagulation and hemostasis. The Sublime and Sublative RF applicators are equivalent to those on the European conformity (CE) marked eLos, eTwo, eMatrix device family. The Matrix Pro applicator utilizes micro-needling technology and is new feature of the Profound Matrix system. The Profound Matrix system, including the Matrix Pro applicator are currently cleared for use in the US under FDA 510k K211217. This study aims to evaluate additional indications for treatment through the electrocoagulation and hemostasis mechanism of action for dermal remodeling and improvement in skin conditions to provide study subjects with a safe and effective alternative treatment that can be performed with minimal risks and decreased downtime. Eligible subjects would be healthy adult volunteers between 18 to 75 years of age seeking clinical treatment for indications as listed above. The research is sponsored by Candela Corporation and planned to be conducted at up to 20 sites globally. From the first subject enrollment to the last subject follow-up, the expected total duration is up to 5 years across all sites. The participants will undergo informed consent, screening and enrollment, treatments for the indication to be treated, and follow-up visits at no cost. The data from this research will assist Candela in optimizing treatment parameters, treatment guidelines, providing input to clinical education and marketing material, and support the research and development of micro-needling technology alongside energy-based devices.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy female and male subjects between 18 to 75 years of age with Fitzpatrick Skin Type I - VI.
2. Willing to receive Profound Matrix treatments with any of the following applicators: Sublime, Sublative RF, and/or Matrix Pro applicator
3. Able and willing to comply with the treatment/follow-up schedule and comply with all study (protocol) requirements.
4. Willing to provide signed, informed consent to participate in the study
5. Willing to have photographs and images taken of the treated areas to be used in evaluations, publications, presentations, and marketing materials (Subject identity will be masked).

Exclusion Criteria:

Any of the following will exclude the subject from the study:

1. Pregnant or planning to become pregnant, having given birth less than 3 months prior to enrollment into the study, and/or breast feeding
2. Pacemaker or internal defibrillator or any active electrical implant anywhere in the body
3. Superficial metal or other implants in the treatment area, except superficial dental implants, unless these implants can be removed or covered with rolled gauze during treatment
4. Skin cancer in the treatment area or history of melanoma
5. History of current cancer and subject has undergone chemotherapy within the last 12 months
6. Severe concurrent conditions, such as cardiac disorders
7. Impaired immune system or use of immunosuppressive medications
8. Herpes Simplex Virus (HSV) in the intended treatment area unless treated following a prophylactic regimen
9. Poorly controlled endocrine disorders such as poorly controlled diabetes
10. Active skin condition in the treatment area such as skin infection, sores, psoriasis, eczema, rash, or open wounds
11. History of abnormal wound healing, keloid, or hypertrophic scar formation, as well as very thin or fragile skin
12. History of collagen vascular disease or vasculitic disorders
13. Known allergy to medication to be used during treatments such as allergy to topical anesthetic (e.g. lidocaine)
14. History of systemic corticosteroid therapy in past six months
15. Tattoos or permanent makeup in the intended treatment area
16. Excessively tanned skin
17. Facelift in the last 12 months
18. Aesthetics treatments/procedures (e.g. facial resurfacing and deep chemical peeling) within the last 4 months within the intended treatment area
19. Neuromodulator injections (e.g. Botox®), collagen, non-permanent dermal filler, or fat injections or other methods of augmentation with injected bio-material in the treated area within the last 3 months
20. Permanent synthetic fillers (e.g. silicone) in the treatment area
21. Absorbable facial threads within the last 1 year or non-absorbable facial threads within the intended treatment area
22. In the opinion of the Investigator, the subject is unwilling or unable to adhere to the study requirements or is otherwise unsuitable for the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2022-05-24 (Actual); Primary Completion 2027-05-24 (Estimated); Study Completion 2028-05-24 (Estimated)

PRIMARY OUTCOMES:
Standardized Clinical Photography | From subject enrollment to completion of 3-month follow-up visit, up to 32 weeks.
  Clinical photography will be taken of treated areas at baseline prior to treatment and all treatment and follow-up visits.
Numerical Rating Scale (NRS) | From the first treatment to the third treatment, up to 16 weeks.
  Subject assessment of treatment discomfort/pain immediately post-treatment via Numerical Rating Scale (NRS). Subjects will be presented a horizontal line scale and asked to make a mark along the scale. Subjects will be asked to rate pain from 0 to 10, with 0 equaling no pain and 10 equaling the worst possible pain. A number is obtained by measuring up to the point the participant has indicated.
Post-treatment Assessment Severity Scale | From the first treatment to the third treatment, up to 16 weeks.
  Skin responses including edema, erythema, pinpoint bleeding, purpura/ecchymosis, petechiae, and microscopic epithelial necrotic debris (MENDs) will be assessed immediately after treatment with a post-treatment assessment severity scale: grade 1 means absent, grade 2 means mild, grade 3 means moderate, and grade 3 means severe.
Investigator Global Aesthetic Improvement Scale (IGAIS) | At 1-month follow-up and 3-month follow-up, up to 14 weeks.
  Investigator Global Aesthetic Improvement Scale (IGAIS) will be assessed at each follow-up visit with score -1 to 3 and corresponding ratings: -1 means worse, 0 means no change, 1 means improved, 2 means much improved, 3 means very much improved.
Subject Satisfaction Scale | At 1-month follow-up and 3-month follow-up, up to 14 weeks.
  Subject satisfaction rating of improvement in indication will be obtained at each follow-up visit. The subject satisfaction scale scores from -2 to 2 with corresponding improvement rate: -2 means very dissatisfied, -1 means somewhat satisfied, 0 means neutral, 1 means somewhat satisfied, 2 means very satisfied.

CONTACTS AND LOCATIONS:
Overall Officials: Konika Schallen, MD, Principal Investigator — Candela Institue for Exellence
Locations (6):
- United States (4):
  - Center for Morden Aesthetic Medicine, Jacksonville, Florida
  - Candela Institue for Excellence, Marlborough, Massachusetts
  - Concierge Medical Arts, Fayetteville, North Carolina
  - Gerrish MedEsthetics, Vienna, Virginia
- Waterfront Skin and Laser, Vancouver, Canada
- Candela European Institue of Excellence, Madrid, Spain